CLINICAL TRIAL: NCT01153048
Title: Randomized Controlled Trial on an Educative Structured Intervention by Peer Educators to Improve HbA1c of Patients With Type 2 Diabetes in the Sikasso Region in Mali
Brief Title: Trial on an Educative Structured Intervention by Peer Educators to Improve HbA1c of Patients With Type 2 Diabetes in the Sikasso Region in Mali
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sante Diabete Mali (Other)
Collaborators: Société Francophone du Diabète (Other); French Development Agency (Other Government); Centre hospitalo-universiaire du Point G de Bamako (CHU Pt G) (Unknown)
Responsible Party: Besançon Stéphane (Program director ONG Santé Diabète Mali), ONG Santé Diabète Mali
Allocation: Randomized | Model: Parallel | Purpose: Supportive Care
Other Study IDs: SDMSFD01
Record Dates: First submitted 2010-06-27; First posted 2010-06-29 (Estimated); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Type 2 Diabetes
Keywords: Intensification of Education; learning nest methodology; peer educators; type 2 diabetes; Mali; the focus of this study is on the intensification of education on the treatment of type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Specific education intervention with peer educators (Experimental)
  Interventions: Other: Intensification of education
- General education session in the health structure (No Intervention)

INTERVENTIONS:
Other: Intensification of education — The main objective is to assess impact of the establishment of involved patients (peer educators) network in Mali. Peer educators and persons targeted by the project will be recruited through Post-Test Club on diabetes (PTC). PTC will be a social support club that provides on going prevention counseling, education and support services to people who have diabetes. PTC represents an important link between patients, educators and general medical services. PTC will be defined as clubs, which are facilitated by well-trained peer educators, and will have 3 objectives: to provide social and emotional support to diabetic patients, to provide assistance in daily management and living with diabetes and to provide linkage to clinical care. To lead the sessions, in clubs, we will use a very innovative methodology for peer education: the learning nests method. To evaluate, we propose a classical randomized controlled experimental (RCT) design, with randomization at the person-level.
  Arms: Specific education intervention with peer educators

SUMMARY:
The main objective is to assess impact of the establishment of involved patients (peer educators) network in Mali. It will be conducted by a multidisciplinary team that brings together high level skills in research projects and in peer education projects. It will be conducted in one country Mali. In the country, it will be completed in one site : the region of Sikasso. This site was chosen because It meet a functional care, access to medicines and a dynamic association of diabetic patients. Peer educators and persons targeted by the project will be recruited through Post-Test Club on diabetes (PTC). PTC will be a social support club that provides on going prevention counseling, education and support services to people who have diabetes. PTC represents an important link between patients, educators and general medical services. PTC will be defined as clubs, which are facilitated by well-trained peer educators, and will have 3 objectives: to provide social and emotional support to diabetic patients, to provide assistance in daily management and living with diabetes and to provide linkage to clinical care. To lead the sessions, in clubs, we will use a very innovative methodology for peer education: the learning nests method. To evaluate, we propose a classical randomized controlled experimental (RCT) design, with randomization at the person-level. For outcome measures, we propose change in HbA1c, increase of social and emotional support and increase of linkage to clinical care. In addition to HbA1c, we propose measuring changes systolic and diastolic blood pressure and weight.

DETAILED DESCRIPTION:
BACKGROUND AND RATIONALE

The World Health Organization (WHO), estimates that the number of people affected by diabetes will rise from 171 million in 2000 to 366 million in 2030, representing a prevalence of 2.8% to 4.4% supposing that obesity will progress. Developing countries will then represent 76% of the world diabetic patients. This growth has justified the alarming report issued by the WHO in 2005 for a rapid mobilization on these new health needs. Access to care, treatment, education and care for complications related to diabetes is a key feature of the resolution passed by the United Nations in December 2006 on diabetes to protect people with diabetes against exclusion situation and increased vulnerability. In developing countries, the explosion of diabetes epidemic and other chronic diseases, is a direct consequence of the widespread emergence of overweight and obesity. For developing countries, the major increase of obesity, which involves both the upper classes that the popular classes, is essentially linked to the emergence of a nutritional transition defined as a gradual change of diets, including a clear increase of fats of animal origin consumption. Finally, the increase of obesity in the southern countries, thus the emergence of chronic diseases like diabetes, is strengthened by the increase of life expectancy and by the growth of physical inactivity.Education on diabetes is known through several names: education of the patient,patient's therapeutic education. All these terms question about the diabetic person's place in a continuous progress involving permanent communication with a care team and the coordination of a care programme. The therapeutic education is more and more becoming a model of care for people with diabetes. Indeed, diabetes is a complex condition, which requires an effective medical management from caregivers and a good autonomous management from the person with diabetes. This dual approach helps to promote choice of healthy lifestyles, improve the quality of life and reduce direct and indirect health costs for society. Educational approaches set up must recognize the critical and fundamental role of psychosocial factors for effective diabetes education. In 1914, Elliott Joslin published a book in which he stressed the importance of training nurses to participate to the education on diabetes and its management [10]. In 1936, insulin appeared and specialized nursing in diabetes had expanded. It became clear that nurses should develop their skills when it comes to education and counselling as well as expertise in clinical care. The publication of the DCCT studies results in 1993 and UKPDS in 1998 amended the diabetes care, from the simple reduction of glycaemia and blood pressure, to the active prevention of complications and in to the intensification of treatment. It was a turning point in the role of diabetes educator. In developed countries, diabetes educators began by considering the key aspects of the insulin doses adaptation, of the changes in eating habits and of the screening for complications, paving the way for the work of specialised nurses and of other caregivers, such as dieticians, chiropodist in diabetes education. Several studies have highlighted, in developed countries, the challenge for health professionals to implement education activities for patients. Above the consideration of the different cultural contexts, the barriers often described by professionals for the establishment of effective patient education are the availability of time and the inadequacy of the initial and continuing training. At hospital, the particular context in which education situations took place do not necessarily encourage the effective setting up of prevention and health practice in every day life. In the context of African health systems that combine low human and financial resources with a very important turn over of staff, it is very difficult to establish specific curricula for diabetes educators, but also to mobilize health staff specifically for this task. In these particular settings, the involvement of peers in the assistance in daily management and living with diabetes, the Social and emotional support and the Linkage to clinical care seems to be a perfect tighten to complement the organization of diabetes care in these countries. The reviews of several studies have shown the very positive results of this approach that can be implemented by following several methodological models. For this study we have chosen to implement and evaluate the impact of the methodology: The Learning Nests approach : Group Education focusing on understanding of key concepts and interactions with social context. This approach developed by health professionals and human sciences seems to be the best suited for the socio economic and cultural contexts which are encountered in Africa. It is based on 5 principles- the building and setting up of learning situations which are based on scientific data of the medical and social/human sciences frame (socioconstructivism, didactic, learning of adults-):

* The integration of the context of life in developing the educational situation
* The work on the operational dimension (use of the knowledge for the action, decision making by the learner), with the support of individual booklets (for the teacher and for the learner)
* The intimate coupling of the educators training and the educational situations for learners
* The implementation in a long-term programme, with precise indicators of results

METHODS

Intended Audience and Setting

Direct beneficiaries in Mali The 150 diabetic patients directly reached by the activities The 7 peer educators trained in the action areas selected in Mali The 30 health agents of the action areas selected in Mali Families and relatives of patients reached by animations in the 2 countries (40000 persons)

Indirect beneficiaries in Mali All the diabetic patients of Mali (3% of the adult population) All the health workers involved in the care of diabetes and NCD in Mali The Malian health systems by improving the monitoring of diabetic patients and reducing complications related to diabetes The Malian population by reducing the risk factors of diabetes and NCD and increasing the quality of life

Indirect beneficiaries in Africa Diabetic patients of French and English speaking African countries which will benefit from the methodology and tools developed Health workers involved in care of diabetes in French and English speaking African countries The health systems and the populations of these countries

General care for diabetes available to Intended Audience

Between 2000 and 2003, many studies have been conducted to identify problems in the prevention and management of diabetes in Africa. These studies have shown similar results:

Health system: the presence of insulin, syringes and testing equipment is vital, but not enough. It must be accompanied by a health system with trained personnel and structures in place. Health systems in Sub-Saharan Africa are organized for the treatment of acute non chronic illnesses. In African countries, the management of diabetes was just available in 2 public structures of the capital. In these structures, the number of consultations was very high and there was no possibility to perform patient education. This situation obliged many patients to do between 500 to 1000 Km to do a diabetes consultation.

Diagnostic: there were problems at all levels with supplies of urine strips, strips for Glucometers, tubes for analyses and reagents. However this was a problem as supplies were expensive.

Education: All studies have shown great difficulty for the implementation of patient education. Indeed, the lack of decentralized consultations made the number of consultation within 3rd reference structures too important for education. The limited human and financial resources also made this education very difficult. In parallel to these problems in the health system, eating habits must be taken into account, for the establishment of adequate education.

Since 2003, Mali and Tanzania have set up advanced programs to improve prevention and diabetes care in 5 parts: research activities / Decentralization of diabetes care / Access to medicine, analysis and medical equipment / support to the creation and setting up of patient associations / primary prevention Training: After the setting up of specific modules with specialized doctors in Mali, 12 diabetes referral doctors were trained in 3 regions of Mali and in 7 communes in the capital Bamako.

Analysis, medical equipment and medicine: each structure, in which referral doctors work, has been equipped with glucometers and urinary strips with a decline of 25 percent of the price on consumables. A several months work with the Central Pharmacy of Mali (PPM) has achieved a national supply and a sharp drop in prices of insulin (actrapide and insulatard), 2 types of diabetes pills (glibenclamide and metformin), measuring strips for ketones and protein in urine, as well as syringes for injections of insulin. These new products have led to a sharp drop in costs for patients (50 percent discount for insulin and division of prices by 10 for diabetes pills). The consultations have also been equipped for the prevention and management of diabetes (measuring apparatus, scale, tensiometer, tuning fork, monofilament, tape measure, registers etc…) Association: the establishment of operational consultations made it possible, month after month, to have decentralized consultations which can take care of a great number of patients. These patients have gradually grouped into association around these consultations.

Primary prevention: wide actions, using the media and community actions, have been implemented to inform and educate people in intervention areas to bring about a change of behaviour in terms of diet, physical activity, but also in the accompanying of patients by the community.

Education: To accompany the care of patients, some first actions have been developed to start an education in health facilities.

For this project we considered it necessary to implement this project in areas where patients have access to equipped quality consultations with availability of testing equipment and medication and strong associations.

Recruitment or approaches to reaching intended audience

A PosT test Club (PTC) will be a social support club that provides on going prevention counseling, education and support services to people who have diabetes. PTC represents an important link between patients, educators and general medical and social economic services.

PTC will be defined as clubs, which are facilitated by well-trained peer educators, and will have 3 objectives:

* To provide social and emotional support to diabetic patients
* To help people feel that they are not isolated and alone with their problems
* To provide a way to meet people and make friends
* To help individual to become more confident and powerful
* To provide a forum to organize activities
* To make links between people from different backgrounds
* To share resources, ideas and information
* To create a public voice which can lead to change To provide assistance in daily management and living with diabetes
* allow patients to appropriate knowledge that is essential to better manage chronic disease.
* allow understanding diabetes and reducing cardiovascular risk by learning how to manage their treatment, diet and regular physical expenditure.
* Patients to stake and analyse the elements of their environment, their representations and ordinary habits with the knowledge coming from the medical field. This analysis of elements in presence should allow everyone to take relevant and appropriate decisions (family, culture, economic, social network).

To provide linkage to clinical care

* Create a network between patients clubs and structures managing diabetes in the action zone
* Define a patient circuit in area where patients clubs will accompany at best patients in structures of care

The intervention areas of the project were selected so that clubs can be established in areas where:

* The consultations for diabetic patients are functional
* Health structures have drugs for care
* Patient associations around consultations are dynamic
* A partnership agreement will be signed between the health authorities, patients' associations and clubs of the area The clubs will be led by educators who are specifically trained diabetic patients. They will be recruited in diabetic patients associations of the area where the club will be located.

The clubs will be made of diabetic patients who will be recruited in diabetes consultations in health facilities and in the diabetic patients association of the area.

Approaches to implementing peer support programs that address the three core components of peer support:

The purpose of this methodology is to set up coordinated training and education activities targeting populations with diabetes based on a pragmatic approach of appropriation and construction of knowledge that takes into account the individual, social, economic, cultural context. This work is being implemented on the basis of group modules specifically designed in their running: are studied the concrete elements of knowledge to mobilize, patients' actions, the role of health professional who is educator, indicators of progress and monitoring during sessions and on the long term. Each patient is gotten to consider the elements involved in his/her disease, and the actions that can be achieved taking into account the feasibility in his/her own context. The education monitoring is envisaged through a data compendium present in the individual books that are given to patients at the end of each education session. The education sessions are built in reference to the socioconstructivist model of learning. Theoretically located, situations are developed with reference to research work coming from different fields: they include the medical dimension (epidemiology, nutrition, endocrinology) and cognitive and social dimension of the chronic disease (learning psychology, sociology of health, Social and medical anthropology). These education sessions allow to work in an effective, assessable and durable way the knowledge coming from the medical sciences (understanding of cardiovascular risk and diabetes, food management, management of physical activity with identification of complications). Patients are gotten to realize their individual potential and social contexts in which they evolve. All the constituent elements of the situation (knowledge, representations of patients, construction of the learning situation) are subject to a detailed analysis that aims to be as objective as possible. By standing out from the prescriptive scheme which structure many education practices, these sessions doubly meet the current needs in therapeutic education: while allowing patients an access to knowledge, they also participate to the establishment of new dynamic in training of health professionals. This approach is therefore proposing a synthesis form, in action of knowledge from various scientific fields. The propositions of understanding and evaluation of the education action impact go beyond the usual practices, as they invest the scope of ordinary habits of patients (which is still insufficiently explored). The animations sessions will allow:

* Patients to appropriate knowledge that is essential to better manage chronic disease.
* Patients to understand diabetes and reduce cardiovascular risk by learning how to manage their treatment, diet and regular physical expenditure.
* Patients to stake and analyse the elements of their environment, their representations and ordinary habits with the knowledge coming from the medical field. This analysis of elements in presence should allow everyone to take relevant and appropriate decisions (family, culture, economic, social network).

In practice the implementation of the methodology takes place in 4 stages:

1. - The training of peer educators who have been identified and recruited to lead the animations
2. - An initial cycle on the themes of knowledge and control of cardiovascular risk (BP, cholesterol, blood sugar, waist measurement, diabetes, treatment and complications). Patients work on modifiable elements influencing health on a vascular viewpoint, identify actions which may have a positive effect on these elements, take into account facts of the real life and choose a realistic action to be done 3- An initial cycle on the subject of food controlling (balance, fat, carbohydrates). Fat intake: analyse and compare foods containing diverse amounts of fats, identify unsaturated and saturated fat content, evaluate and correct the amount of fats in diet if necessary; understand the relation between fats, visceral adiposity, and glycaemia regulation 4- An initial cycle on the themes of physical activity. Exercise: quantify his/her own actual physical activity on a weekly basis, compare to recommendations, analyse conditions and feasibility of implementing it in real life.

In the frame of these 3 Education sessions, patients are required to:

* Analyse knowledge that appear in various forms, including forms tailored to illiterate and uneducated patients (colour codes, presence of photographs)
* Act on knowledge: the patient observes, makes hypothesis, tests, compare, infer, analyses and makes connections.
* Interact with other learner, which gives education its social dimension.

During each education session, interactive workshops will allow to work on: a balanced diet, carbohydrates in the diet, cardiovascular risk and understanding of diabetes. For each situation, a one-day training will be conducted by trained peer educators with theoretical input on the issue dealt with, put in practice situation, analyses of issues outside the framework and put in "safety education". These training days will be implemented with 8-10 patients (1H 30) and 3 meetings will take place over a period of 2 to 3 months. The educational booklets will be available for patients at the end of the meeting.

The implementation of this comprehensive methodology, including the selection of action areas, the recruitment of educators as well as patients and the implementation of education through the learning nests, will allow a support by:

1. - Assistance in daily management and living with diabetes : the provision for patients of supports understandable and discussed in situation facilitates the appropriation of knowledge over time: the written materials are discovered, approached and negotiated in situation, with the help of the educator. The patient takes the written materials at home, and keeps them carefully for the possibility of organizing the monitoring and the daily management of his diabetes and his life over the long term.
2. - Social and emotional support: the methodology of patients and educators recruitment through patients' associations and educational clubs will provide a very strong social and emotional support to patients. The group education methodology will also allow patients to support each other. Indeed, the work in interaction with other students, gives education a dimension allowing a very strong emotional support. The possibility of keeping the written material negotiated and worked in situation (booklets), will disseminate information within the family or/and in the social network of the trained patient (without risk of knowledge transformation, as the booklet is a reference). This possibility increases the number of people informed on the prevention of chronic diseases, prevention of complications but also allow bringing the necessary information to the family and social network of the formed patient which will strengthen the social and emotional support brought to the patient.
3. - Linkage to clinical care: The choice of intervention areas for Mali and Tanzania has been done taking into account the areas where the care of patients is complete with: an effective and operational diabetes consultation, medicines available and a dynamic diabetic patients association. In these areas, the approach is integrated. The addition of the education methodology by the educators will represent another step in the care pyramid of diabetes. All health workers of the area will be involved in the implementing and monitoring of the process. In addition to the role of educator, educators will also be trained to accompany patients in health facilities that manage diabetes in the intervention area. All peer educators will receive a tool representing the circuit of the patient in the intervention area and will give them to each patient during the animations. Finally, after the meetings patients may accompany each other in the health system.

Approaches to evaluation

Experimental Design. we would like to propose a specific evaluation design and endpoint measures for our study site. We propose a classical randomized controlled experimental (RCT) design, with randomization at the person-level following recruitment, informed consent, and the collection of baseline data. Given the potential value of peer support to the 240 million persons worldwide with diabetes, the large majority of whom do NOT live in industrialized countries [30 ], it would be tragic to waste the opportunity to evaluate peer support in Africa by using a design that is not immediately convincing to all concerned, including the donor agencies and nations who will be asked to fund much of the future roll-out of peer support but may be quite suspicious of "evidence" from would-be aid recipients. Widespread recognition of our results by donors and African leaders and clinicians, which can only come from publication in a global journal like Lancet or BMJ or PLOS Medicine, also requires the strongest possible experimental design.

The RCT design provides the greatest possible internal validity and we see no reasonable alternative to it in our setting. A person-level randomized design is also surprisingly feasible in Mali. In these locations we have already achieved a well-functioning clinical system for diabetes care that can achieve guideline-adherent care (based on African regional diabetes guidelines and IDF guidelines for poor and developing countries). Therefore, the next step, the introduction of peer support programs, can be accomplished without inducing significant cross-contamination; that is, the creation of peer support groups will not cause major changes in the health care delivery process that will spill over to control-group subjects. Moreover, because face-time with physicians and physician-extenders is so limited in impoverished settings like ours, we do not foresee much scope for physicians (who cannot be blinded to experimental assignment) to change the treatment of controls in a compensatory way. However, to prevent this we will train all the relevant caregivers in the importance of maintaining experimental separation, and we will track all diabetes-related treatments to detect any biases that might emerge.

Outcome Measures. We propose change in HbA1c as the primary study measure because (a) it is a "hard" measure that is not subject to short-term variability or to the social-desirability bias that can influence self-reported data; (b) it responds directly to the full breadth of the behaviors that peer-support intends to modify, from diet and exercise to self-glucose monitoring to proper use of medications; and (c) it is the physiologic parameter that is most urgent for persons with diabetes to improve. In addition to HbA1c, we also propose measuring changes systolic and diastolic blood pressure, and weight.

Method for the randomization Patients will be selected in the list of diabetic patients followed in the two consultations diabetes in Sikasso.

From this numbered list a lottery will be conducted through a random number table to constitute the intervention group. From this numbered list a lottery will be conducted through a random number table to constitute the control group. We will verify that all patients randomly selected to form these groups meet the criteria inclusion of groups (see below). The randomization list will be kept by the principal investigator of the survey.

Calculation of the size of study

In this trial, patients were randomized into 2 groups:

* Group 1: Intervention educational peer group associated with the traditional education
* Group 2: classic education without intervention with peer education

It is assumed that in the reference group, the value of HbA1c was 8.5% with a correct standard deviation of 1.5, to correct (previous study conducted in the framework of the NGO Health Diabetes Mali underway published) and we consider that the strategy would be interesting if the assessed value of the mean HbA1c decreased by 1 percentage point HbA1c and standard deviation of 0.5 ..

In this situation, with a risk α of 5% and power 1-β of 80%, it must include 60 patients in each group. To reflect a proportion of patients lost to follow up to 20%, we decided recruit 75 patients per group were 150 patients in total

Eligibility criteria The study will be conducted among patients with type 2 diabetes followed in the decentralized units of the city of Sikasso (third administrative region of Mali). The methodology of choice for patients is described in the paragraph above. The recruitment will be held during the months of June-July 2010.

Inclusion Criteria

* Patients treated in units diabetes in the intervention area and performing regularly consultations
* Patients with type 2 diabetic insulin-treated or untreated
* Poorly controlled diabetes with HbA1c ≥ 8%
* Patients who agreed to undergo the whole process of peer education
* Patients who agreed to carry out all biological measures included in the Protocol
* Patients aged 30-80 years

Criteria for non-inclusion

* Diabetic patients not performing their monitoring units in the area of diabetes intervention
* Patients with diabetes followed in units of the intervention area but not performing regular their consultations
* Patients with type 1 diabetes
* Scalable severe complications within 3 months preceding infection, complications heart disease, severe renal
* Associated diseases threatening or vital functional
* Refusal to participate in the study

Data management and analysis

Data Management. We propose to require that study data be entered and verified (re-entered) from study sites via the internet, as we are currently doing in our multi-country study of the impact of diabetes, using an SQL interface that meshes with EPI-Info. By providing unique field numbers for each response-item, comparability can be maintained despite translations of text and more substantive variations that might be required from site to site. Web-based data entry can now be accomplished even from towns in Africa and we will do this for our own data even if a program-wide web-based data entry system is not developed. . We propose to store the hard copies of study forms in locked cabinets under the control of the PIs in Bamako, Mali.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated in units diabetes in the intervention area and performing regularly consultations
* Patients with type 2 diabetic insulin-treated or untreated
* Poorly controlled diabetes with HbA1c ≥ 8%
* Patients who agreed to undergo the whole process of peer education
* Patients who agreed to carry out all biological measures included in the Protocol
* Patients aged 30-80 years

Exclusion Criteria:

* Diabetic patients not performing their monitoring units in the area of diabetes intervention
* Patients with diabetes followed in units of the intervention area but not performing regular their consultations
* Patients with type 1 diabetes
* Scalable severe complications within 3 months preceding infection, complications heart disease, severe renal
* Associated diseases threatening or vital functional
* Refusal to participate in the study

Ages: 30 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2010-06 (Actual); Primary Completion 2011-07 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
compare the improvement of HbA1c 1 year after an intervention led by peer educators, versus a conventional care in health centre

SECONDARY OUTCOMES:
Study the evolution of bio clinical parameters: fasting glucose, weight, BMI, blood pressure, waist size

CONTACTS AND LOCATIONS:
Locations (1):
- ONG Santé Diabète Mali, Bamako, Mali